CLINICAL TRIAL: NCT00031343
Title: A Randomized, Controlled Study to Assess the Impact of Highly Active Antiretroviral Therapy to Hepatitis C Therapy in Patients Coinfected With HIV-1 and Treated With Peginterferon Alpha-2b and Ribavirin
Brief Title: The Impact of HAART on Response to Hepatitis C Treatment in Patients Taking Peginterferon Alpha-2b and Ribavirin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020139; 02-I-0139
Record Dates: First submitted 2002-03-02; First posted 2002-03-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-04

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Liver Disease; Virologic Response; Immune Mechanisms; Eradication; Antiviral Therapy; HIV; Hepatitis C; HCV; Coinfection
MeSH Terms: conditions — HIV Infections; Hepatitis C; Liver Diseases; Coinfection | interventions — Antiretroviral Therapy, Highly Active

INTERVENTIONS:
Drug: highly active antiretroviral therapy (HAART)

SUMMARY:
This study will evaluate how controlling HIV infection with HAART (highly active antiretroviral therapy) affects the response to hepatitis C treatment with peginterferon alpha-2b and ribavirin in HIV-infected patients with chronic hepatitis C. HIV worsens liver disease caused by hepatitis C. Since treatment of HIV infection with HAART improves immune function, it may be beneficial to start HAART before treating HCV.

HIV-infected patients 18 years of age and older with chronic hepatitis C infection may be eligible for this study. Patients must have an HCV viral load greater than 2000 copies/mL and a CD4 count that is either more than 500 cells/mm3, or more than 350 cells/mm3 with an HIV viral load no greater than 40,000 particles/mL. Candidates will be screened for current or previous diseases, conditions or treatments that may exclude them from this study. Screening includes a medical history and physical examination, eye examination, blood and urine tests, chest X-ray, electrocardiogram (EKG), liver ultrasound, and, possibly, a liver biopsy, if a recent one is not available. The liver biopsy is optional and is done to determine the severity of liver disease. Patients will be sedated for this test. The skin in the area over the biopsy site is numbed with a local anesthetic, and a needle is inserted rapidly into and out of the liver to obtain a small tissue sample. Patients remain in the hospital overnight for monitoring. Women of childbearing age will have a pregnancy test.

Patients enrolled in the study will be randomly assigned to one of the following treatment groups: 1) pegylated interferon and ribavirin for 48 weeks (control group); or 2) HAART for 6 months, followed by 48 weeks of pegylated interferon and ribavirin.

HAART group - Patients taking HAART will be followed in the clinic every 2 weeks for the first month and then monthly for the next 5 months. After 6 months of HAART they will begin taking pegylated interferon and ribavirin and will follow the dosing and follow-up schedule outlined below for patients in the control group.

Control group - Patients will have weekly injections under the skin of peginterferon alpha-2b and ribavirin pills daily by mouth. Clinic visits will be scheduled as follows:

* Days 1, 3, 7, and 21 - Blood will be drawn for safety tests and to measure blood levels of HIV and HCV. HCV medications will be injected on days 7 and 21.
* Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 52, 56, and 64 - Blood and urine tests will be done to determine the side effects of pegylated interferon and ribavirin treatment and its effect on the HCV infection. Eye examinations will be done every 3 months.
* Week 48 or end of treatment - Treatment with pegylated interferon and ribavirin will stop after 48 weeks. At this time (or earlier for those who do not complete the 48 weeks of treatment), patients will return to the clinic for a routine visit, blood tests (including a test for hepatitis B) and abdominal ultrasound. Patients may also be hospitalized for 2 days for a repeat optional liver biopsy.
* Week 72 and extended follow-up visits - At week 72, patients will return for blood tests and a routine clinic visit. HCV viral load will be measured. Follow-up visits every 3 months for an additional year will include a blood test to measure HCV viral load and a complete physical examination.

DETAILED DESCRIPTION:
Coinfection with the human immunodeficiency virus (HIV) and the hepatitis C virus (HCV) has risen dramatically since the explosion of the HIV pandemic twenty years ago, with one third of all HIV positive persons also infected with HCV. Numerous studies have suggested that HIV exacerbates several steps in the natural history of hepatitis C, and as survival among HIV-infected patients increases, hepatitis C-related morbidity and mortality is expected to follow a similar trend in coinfected patients. Some investigators advocate the initiation of highly active antiretroviral therapy (HAART) for this population prior to the initiation of HCV therapy. It is postulated that HAART will improve the host immune function by increasing the CD4+ cell count and decreasing HIV viral load, thought to be advantageous for patients starting HCV therapy. Despite its promising hypothesis, whether HAART ultimately leads to a reduction in HCV load in coinfected persons remains controversial. This is a non-blinded, randomized controlled trial to evaluate the impact of HAART on the immunologic, virologic, and clinical responses to HCV treatment with peginterferon and ribavirin in coinfected individuals with CD4 greater than or equal to 500 cells/mm (3) or greater than or equal to 350 cells/mm(3) and a viral load less than or equal to 40,000 copies/mL. The study will also address the safety and efficacy of administering a combination of HAART along with peginterferon alpha-2b and ribavirin to HIV-infected individuals. 128 patients who are coinfected with HIV and HCV will be recruited for the study and randomized to receive one of two treatment regimens: 1) control group: will be treated with peginterferon alpha-2b and ribavirin for 48 weeks, or 2) experimental group: will be treated with highly active antiretroviral therapy for six months. At that point, they will begin receiving peginterferon alpha-2b and ribavirin at the same doses as the control group for 48 weeks. During the 72-week follow up period, these patients will be monitored for both HCV and HIV viral loads and CD4+ lymphocyte counts. The results of the study will enable us to better delineate the relationship between the immune reconstitution effects induced by HAART and the clinical, immunologic, and virologic responses of coinfected persons treated with peginterferon and ribavirin. In addition, evaluating the safety of coadministering peginterferon, ribavirin, and HAART will further refine the best therapeutic regimen for this patient population.

ELIGIBILITY:
INCLUSION CRITERIA:

Age greater than or equal to 18 years

Documentation of HIV-1 infection by a licensed ELISA test and confirmed by a Western Blot

CD4 greater than or equal to 500 cells/mm(3) or CD4 greater than or equal to 350 cells/mm(3) and HIV VL less than or equal to 40,000 copies per milliliter

CD4 nadir not below 200 cells/mm(3)

If not HAART naive, history of HIV VL suppression while on HAART treatment.

Patients who are currently on HAART but do not meet criteria for the initiation of HAART according to current DHHS guidelines must be willing to come off their regimen 3 months prior to study initiation.

Documentation of Hepatitis C infection by demonstration of a positive test for hepatitis C antibody.

HCV RNA level greater than 2000 copies per milliliter by polymerase chain reaction

Patients naive to HCV treatment at time of enrollment.

Serum creatinine less than or equal to 1.5 mg/dL

Serum phosphorus greater than or equal to 2.2 mg/dL (normal range NIH 2.3-4.3 mg/dL)

Neutrophil count greater than or equal to 1000 cells/mm(3)

Platelets greater than or equal to 75,000/mm(3)

Hemoglobin greater than or equal to 8.0 mg/dL

ALT less than 7 X the NIH upper limit of normal

Not pregnant or breast-feeding. Pregnancy tests must be negative within two weeks prior to dosing with study medications.

Due to the teratogenic effects of ribavirin, for women of child-bearing age, the use of effective contraception during the study will be required. These include abstinence, surgical sterilization of either partner, barrier methods such as a diaphragm, condom, cap or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter the metabolism of hormonal contraception.

Patients must have a primary MD responsible for their HIV infection and liver disease.

Willing to designate a person for durable power of attorney on NIH form for medical research and medical care purposes at the NIH Clinical Center.

Ability to learn how to safely inject medication subcutaneously or have a family member, relative or partner who is willing to learn to inject study medication.

Competency to sign informed consent and willingness to comply with study requirements and clinic policies.

Willingness to have blood and tissue specimens stored in NIH facilities.

Child-Pugh score less than 6.

Willingness for female patients to practice at least two reliable forms of effective contraception during treatment with ribavirin. Effective means of contraception include barrier and hormonal methods.

Willingness for male patients to practice effective contraception during treatment with ribavirin, including barrier methods.

EXCLUSION CRITERIA:

PT-INR (in the absence of anti-cardiolipin Ab) by greater than or equal to 2.

Organ transplant recipient

Recent HIV seroconverters (must be 6 months or more with documented HIV diagnosis).

Patients who are medically indicated to begin HAART therapy

Elevated alpha-fetoprotein level (greater than or equal to 100 ng/mL).

Coexisting neoplastic disease requiring cytotoxic therapy.

Have had cancer other than Kaposi's sarcoma of the skin, other skin cancers treated by resection, Bowen's disease, or localized cervical or anal cancer in the 5 years prior to enrollment

Have had significant renal dysfunction within the previous 12 months or evidence of significant protein wasting

Severe cardiac or pulmonary decompensation as assessed by the PI.

Severe liver decompensation or advanced cirrhosis patients

Severe psychiatric disorder that would interfere with the adherence to protocol requirements.

Autoimmune disorders including inflammatory bowel diseases, and optic neuritis as assessed by the PI.

Uncontrolled seizure disorder

Severe retinopathy.

Direct bilirubin more than or equal to 2 times ULN.

No patients using long-term systemic corticosteroids, immunosuppressives, IL-2, or cytotoxic agents within 60 days of enrollment.

Active systemic infections (other than hepatitis C and HIV).

Liver disease caused by reasons other than hepatitis C like HBV, HDV, Wilson's hemochromatosis, or autoimmune hepatitis (ANA greater than or equal to 3.0) except history of drug-associated hepatitis with discontinuation of the causative agent.

Hepatic mass suggestive of hepatocellular carcinoma.

Current alcohol or substance use.

Any systemic illness that will make it unlikely that the subject will be able to return to NIH for the required study visits.

Evidence of gastrointestinal malabsorption, chronic nausea, or vomiting

Any pre-existing hemoglobinopathy.

Patients taking any of the following medications: rifampin/rifampicin, rifabutin, pyrazinamide, isoniazid, ganciclovir, thalidomide, oxymetholone, immunomodulatory treatments (including supraphysiologic doses of steroids and radiation, and antineoplastic agents).

Patients taking any investigational drugs and herbal remedies, and other complementary/alternative medications for possible or perceived effects against HCV.

Patients cannot be receiving IL-2 during participation in this study.

Ribavirin is contraindicated in male partners of women who are pregnant. Therefore, potential male patients with pregnant female partners will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128
Dates: Start 2002-02; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] National Institutes of Health Consensus Development Conference Panel statement: management of hepatitis C. Hepatology. 1997 Sep;26(3 Suppl 1):2S-10S. doi: 10.1002/hep.510260701. PMID 9305656
- [Background] Alter MJ, Mast EE. The epidemiology of viral hepatitis in the United States. Gastroenterol Clin North Am. 1994 Sep;23(3):437-55. PMID 7989088
- [Background] Alter MJ, Margolis HS, Krawczynski K, Judson FN, Mares A, Alexander WJ, Hu PY, Miller JK, Gerber MA, Sampliner RE, et al. The natural history of community-acquired hepatitis C in the United States. The Sentinel Counties Chronic non-A, non-B Hepatitis Study Team. N Engl J Med. 1992 Dec 31;327(27):1899-905. doi: 10.1056/NEJM199212313272702. PMID 1280771